CLINICAL TRIAL: NCT07124429
Title: A Comparative Evaluation of the Effects of Reformer Pilates and Standard Physiotherapy on Rehabilitation After Femoral Lengthening Surgery.
Brief Title: Effects of Reformer Pilates and Standard Physiotherapy on Rehabilitation After Femoral Lengthening Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6683
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Femur; Short
Keywords: femur
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates (Experimental): Reformer Pilates
  Interventions: Other: Reformer Pilates
- conservative treatment (Active Comparator): conservative treatment
  Interventions: Other: conservative treatment

INTERVENTIONS:
Other: Reformer Pilates — Reformer pilates is a form of exercise that uses a specialized machine with a sliding carriage and springs to provide resistance. It is highly effective for improving core strength, flexibility, and muscle tone while also promoting better posture and balance.
  Arms: Reformer Pilates
Other: conservative treatment — Conservative physiotherapy is a treatment approach that aims to manage pain and improve function using non-surgical methods. This treatment often includes methods like applying hot packs to relax muscles and increase circulation, and using a TENS (Transcutaneous Electrical Nerve Stimulation) device to help relieve pain.
  Arms: conservative treatment

SUMMARY:
The femur, which forms the foundation of the lower extremity's skeletal system, is one of the most critical bones in the human body due to both its structural integrity and its functional duties.

DETAILED DESCRIPTION:
Surgical interventions aimed at correcting femur length have held a very important place in the development of orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 45 years
* Male gender
* Having undergone bilateral femoral lengthening surgery for cosmetic purposes only
* The lengthening operation having been performed solely with the LON technique

Exclusion Criteria

* Female patients
* Patients who have undergone unilateral femoral lengthening surgery
* Patients under 18 or over 45 years of age

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-11 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Muscle strength assessments | 8 weeks
  Muscle strength assessments were performed using a MicroFET brand handheld dynamometer.
Muscle shortness | 8 weeks
  Muscle shortness was measured using standard clinical evaluation methods. The quadriceps femoris and hamstring muscles are major opposing groups in the thigh, while the tensor fasciae latae (TFL) is a key muscle involved in hip movements.
Joint Range of Motion | 8 weeks
  Joint range of motion measurements were evaluated separately for the right and left sides using a standard goniometer
Muscle Reaction Time | 8 weeks
  The BlazePod TTM (Play Coyotta Ltd.) device was used for the assessment of muscle reaction time. This device is a wireless system consisting of LED lights and a central controller, and it's designed to measure a participant's response time to specific light signals.
Daily Living Activities | 8 weeks
  Functional status was assessed using the Barthel Activities of Daily Living Index, which ranges from 0 (total dependence) to 100 (complete independence), with higher scores indicating a better outcome.
Pain Assessment | 8 weeks
  Participants' pain levels were evaluated using the Visual Analog Scale (VAS). All data was collected by a physiotherapist in a one-on-one session within a clinical setting and manually recorded on standard evaluation forms.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahceşehir University Health Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No